CLINICAL TRIAL: NCT06434077
Title: Clinical Trial Protocol: Randomized Placebo-Controlled Pilot Study of GcMAF (Soloways TM) in Patients With Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW011
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; GcMAF (Gc Macrophage Activating Factor); Nagalase; Inflammation Markers; Response Evaluation Criteria in Solid Tumors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGMAF group (Experimental): GcMAF injections (100 ng)
  Interventions: Biological: GcMAF injections (100 ng)
- placebo group (Placebo Comparator): placebo injections (100 ng)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: GcMAF injections (100 ng) — The GcMAF 100 ng (Gc protein macrophage-activating factor) will be injected subcutaneously.
  Arms: CGMAF group
Other: placebo — the placebo solution will be injected subcutaneously 100 ng.
  Arms: placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled pilot study aims to evaluate the efficacy and safety of GcMAF in reducing nagalase levels and improving clinical outcomes in female patients with metastatic breast cancer over six months. Sixty patients will be randomized into two groups receiving either weekly GcMAF or placebo injections. The primary endpoint is the change in serum nagalase levels from baseline to six months. Secondary endpoints include clinical status, quality of life, adverse effects, and markers of inflammation and immune activity. Tumor response will be assessed using RECIST criteria, and quality of life will be measured with the EORTC QLQ-C30 questionnaire. Immune and inflammation markers will be evaluated using flow cytometry and ELISA. Adverse events will be monitored and categorized according to severity. Inclusion criteria include confirmed metastatic breast cancer, completion of one line of systemic therapy, adequate organ function, and elevated serum nagalase levels. The study will involve baseline measurements, monthly assessments, and final evaluations to compare changes in nagalase levels and other clinical outcomes between the GcMAF and placebo groups.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled pilot study aims to evaluate the efficacy and safety of GcMAF (Gc Macrophage Activating Factor) in female patients with metastatic breast cancer. The primary objective is to assess the reduction in serum nagalase levels, an enzyme associated with tumor activity, over a six-month period, and to evaluate improvements in clinical outcomes. The study involves 60 patients who will be divided into two groups: one receiving weekly injections of GcMAF and the other receiving a placebo.

Patients eligible for the study must have histologically or cytologically confirmed metastatic breast cancer, completed at least one line of systemic therapy, and have elevated serum nagalase levels. Additional inclusion criteria include female patients aged 18 to 70 years, ECOG performance status of 0 to 2, adequate bone marrow, liver, and renal function, and an estimated life expectancy of at least six months. Patients must also agree to use effective contraception and provide informed consent.

The primary endpoint is the change in serum nagalase levels from baseline to six months. Measurements will be taken at baseline, monthly, and at the end of the study using standardized enzymatic assays. Secondary endpoints include clinical status, assessed through objective tumor response using RECIST criteria and performance status using the ECOG scale, quality of life evaluated through EORTC QLQ-C30 questionnaires, immune activity measured by flow cytometry for various immune cell subsets, and inflammation markers such as CRP, interleukins, and TNF-alpha measured by ELISA. Adverse effects will be monitored weekly and categorized according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

The study procedures include initial screening to measure baseline nagalase levels and assess eligibility, followed by randomization into the GcMAF or placebo groups. Patients will receive weekly injections for six months, with monthly assessments of nagalase levels, clinical status, quality of life, and blood samples for immune and inflammation markers. Interim assessments will occur at three months, with final assessments and data analysis at six months.

Exclusion criteria include the presence of other active malignancies, severe uncontrolled illnesses, pregnancy or breastfeeding, previous treatment with GcMAF, and known hypersensitivity to the study drug components. The study timeline consists of patient recruitment and baseline measurements in the first month, followed by six months of treatment and monitoring, with interim and final assessments and subsequent data analysis.

This study aims to determine if GcMAF can significantly reduce serum nagalase levels and improve clinical outcomes, including tumor response, performance status, quality of life, and immune and inflammation markers, in patients with metastatic breast cancer. The results will provide insight into the potential therapeutic benefits of GcMAF for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Histologically or cytologically confirmed metastatic breast cancer.
  * Evidence of metastatic disease, confirmed by imaging studies (CT, MRI, or PET scans) and/or biopsy. 2. Prior Treatment:
  * Patients must have completed at least one line of systemic therapy (e.g., chemotherapy, hormone therapy, targeted therapy) for metastatic breast cancer.
  * A minimum of 4 weeks must have elapsed since the last chemotherapy, targeted therapy, or radiotherapy before starting the study treatment. 3. Age:
  * Female patients aged 18 to 70 years. 4. Performance Status:
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2. 5. Life Expectancy:
  * Estimated life expectancy of at least 6 months. 6. Laboratory Values:
  * Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, and hemoglobin ≥ 9 g/dL.
  * Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver metastases).
  * Adequate renal function: Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60 mL/min/1.73 m^2 (calculated using the Cockcroft-Gault formula). 7. Contraception:
  * Women of childbearing potential must agree to use effective contraception (e.g., hormonal contraceptives, intrauterine device, barrier methods, or abstinence) during the study and for at least 6 months after the last dose of study treatment. 8. Informed Consent:
  * Ability to understand and willingness to sign a written informed consent document.

    9. Compliance:
  * Willingness and ability to comply with the study protocol, including scheduled visits, treatment plans, laboratory tests, and other study procedures. 10. Nagalase Levels: • Elevated serum nagalase levels above the normal range, indicating active tumor burden.

Exclusion Criteria:

* Concurrent Malignancies:

  * Presence of other active malignancies (excluding adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix). 2. Severe Comorbid Conditions:
  * Severe uncontrolled concurrent illness, such as significant cardiovascular disease (e.g., uncontrolled hypertension, recent myocardial infarction), severe pulmonary conditions (e.g., uncontrolled asthma, chronic obstructive pulmonary disease), or active infections requiring systemic therapy. 3. Pregnancy and Lactation:
  * Pregnant or breastfeeding women. 4. Previous GcMAF Treatment:
  * Previous treatment with GcMAF. 5. Allergies and Sensitivities:
  * Known hypersensitivity to any component of the study drug or its formulation.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Nagalase Levels | 6 months

SECONDARY OUTCOMES:
Change in RECIST (Response Evaluation Criteria in Solid Tumors) criteria. | 6 months
MRI changes in cancer volume | 6 months
Tumor response | 6 months
  one of 4 categories Complete Response (CR), Partial Response (PR), Stable Disease (SD),Progressive Disease (PD)
Eastern Cooperative Oncology Group (ECOG) performance status change | 6 months
EORTC QLQ-C30 change | 6 months
  (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire
CD4+T cells percentage | 6 months
CD8+T cells percentage | 6 months
NK cells percentage | 6 months
CRP percentage | 6 months
IL-6 percentage | 6 months
IL-10 percentage | 6 months
tumor necrosis factor-alpha (TNF-α) necrosis factor-alpha (TNF-α) | 6 months
Adverse events | 6 months
  any adverse events will be reported
rank of adverse event severity in numbers | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia